CLINICAL TRIAL: NCT06655389
Title: Correlation Between PLA Levels and Disease Severity in Patients With Sepsis Cardiac Insufficiency
Status: Recruiting | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Xiu Shengyao, physician, Dongzhimen Hospital, Beijing
Other Study IDs: Nan Guo（Dongzhimen）
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Sepsis Cardiac Insufficiency
Keywords: Sepsis cardiac insufficiency; PLA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis cardiac insufficiency group: Cardiac dysfunction or hemodynamic abnormalities in patients with sepsis, combined with abnormal cardiac ultrasound findings, markers of myocardial injury, and/or markers of cardiac function
  1. From April 2024 to December 2026, in the first ICU area of Dongzhimen Hospital, Beijing University of Chinese Medicine,Hospitalized patients in Zone II;
  2. consistent with the diagnosis of sepsis cardiac insufficiency;
  3. Age ≥ 50 and ≤ 90 years old;
  4. SOFA score≥ 2 points;
  5. Within 24 hours of the diagnosis of cardiac insufficiency in sepsis;
  6. The patient or his/her family members sign the informed consent form.
- Healthy subjects: 1. Aged ≥ 50 and ≤ 90 years old, permanent residents of Beijing community;
  2. Good health (blood routine, liver and kidney function, blood lipids, blood coagulation, no obvious abnormalities, no diagnosis cardiac insufficiency, acute coronary syndrome, old myocardial infarction, or cardiomyopathy);
  3. There is no history of long-term use of drugs that affect platelet function and coagulation function, and those who are willing to cooperate with the test Crowd;
  4. The subject himself signed the informed consent form.

SUMMARY:
Sepsis cardiac insufficiency is characterized by high morbidity and mortality. Studies have shown an association between elevated PLA levels in patients with sepsis and clinical outcomes of cardiac dysfunction. This study will explore the correlation between circulating PLA levels and organ dysfunction and disease severity in SIMD patients in the form of a cross-sectional study.

DETAILED DESCRIPTION:
Sepsis cardiac insufficiency is an unsolved problem in the field of severe disease, which is characterized by high morbidity and high mortality. Several studies have found that infectious factors activate platelets and inflammatory cells, damage the vascular endothelium, and cause leukocytes to interact with platelets to form platelet-leukocyte aggregates, and elevated PLA levels in patients with sepsis are associated with the clinical outcome of cardiac dysfunction. The literature studies have shown that the serum PLA level in sepsis patients is significantly increased, and the PLA level is positively correlated with the severity of cardiac dysfunction in sepsis patients, and the formation of PLA is regulated by the binding of CD62P on the surface of activated platelets and PSGL-1 on the surface of leukocytes. This study will explore the correlation between circulating PLA levels and organ dysfunction and disease severity in patients with SIMD in the form of a cross-sectional study, in order to provide a new potential direction for the evaluation and treatment of SIMD.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis cardiac insufficiency group

  1. From April 2024 to December 2026, in the first ICU area of Dongzhimen Hospital, Beijing University of Chinese Medicine, Hospitalized patients in Zone II;
  2. consistent with the diagnosis of sepsis cardiac insufficiency;
  3. Age ≥ 50 and ≤ 90 years old;
  4. SOFA score≥ 2 points;
  5. Within 24 hours of the diagnosis of cardiac insufficiency in sepsis;
  6. The patient or his/her family members sign the informed consent form. Healthy subjects

  <!-- -->

  1. Aged ≥ 50 and ≤ 90 years old, permanent residents of Beijing community;
  2. Good health (blood routine, liver and kidney function, blood lipids, blood coagulation, no obvious abnormalities, no diagnosis cardiac insufficiency, acute coronary syndrome, old myocardial infarction, or cardiomyopathy);
  3. There is no history of long-term use of drugs that affect platelet function and coagulation function, and those who are willing to cooperate with the test Crowd;
  4. The subject himself signed the informed consent form.

Exclusion Criteria:

* 1) Diagnosed with acute coronary syndrome, old myocardial infarction, and coronary heart disease revascularization of patients; (2) Cardiac insufficiency due to cardiomyopathy, such as hypertrophic cardiomyopathy, dilated cardiomyopathy, myocardial amyloidosis, diabetic cardiomyopathy, hypothyroidic cardiomyopathy, etc.; (3) Due to heart knots Cardiac insufficiency caused by structural abnormalities, arrhythmias, cor pulmonale, nephroheart syndrome, etc.; (4) Impact Survival of severe primary diseases, including: uncontrolled malignant tumors that have metastasized in multiple places and cannot be resected, and blood disease, novel coronavirus infection and HIV, etc.; (5) Liver and kidney dysfunction with a single SOFA score of ≥3 points in liver or kidney handicappers; (6) Those who have been continuously using immunosuppressants or organ transplantation in the past 6 months; (7) 7 consecutive days prior to enrollment Those who have used corticosteroids, converted to methylprednisolone dose≥ 20mg/day; (8) Pregnant and lactating women; (9) Take or Injection of drugs that affect platelet function and coagulation function; (10) Those who have participated in other clinical trials within 30 days.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Comparison of patients with sepsis cardiac insufficiency with healthy people
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PLA | At the time of admission
  Platelet-leukocyte aggregate levels

SECONDARY OUTCOMES:
Echocardiography | At the time of admission
  Echocardiography assesses cardiac function
APACHEII | At the time of admission
  Acute Physiology and Chronic Health Evaluation
SOPA | At the time of admission
  Sequential organ failure score
BNP | At the time of admission
  Brain natriuretic peptide

CONTACTS AND LOCATIONS:
Overall Officials: Nan Guo, Chief physician, Principal Investigator — DongzhimenH，Beijing
Locations (1):
- DongzhimenH，Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No